CLINICAL TRIAL: NCT05217290
Title: The Effect of Health Education Given to Prediabetes Patients by Videoconferencing on Self-management and Exercise
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Melek ÖZTÜRK, lecturer, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HASANKU_MELEKO
Record Dates: First submitted 2021-09-07; First posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: PreDiabetes
MeSH Terms: conditions — Prediabetic State | interventions — Transtheoretical Model

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experiment group (Experimental)
  Interventions: Behavioral: transtheoretical model
- control group (No Intervention)

INTERVENTIONS:
Behavioral: transtheoretical model — The Transtheoretic Model is a conscious behavior change model and argues that behavior change is a process and that the attempts made in accordance with the change stage of the individual facilitate the change, otherwise resistance to behavior change is developed.
  Arms: experiment group

SUMMARY:
The research will be carried out in order to investigate the effect of health education given to prediabetes patients by video conference method on self-management and exercise.

The work will be carried out in two stages. In the first stage, the validity and reliability study of the Scale for Process of Exercise Engagement (SPEE) that was developed on prediabetes patients will be conducted and the scale will be adapted to the Turkish society. In the second stage, the effect of health education, which was prepared on the basis of the Transtheoretic Model and will be given by video conferencing, on the exercise status of prediabetes patients, on hunger, postprandial blood sugar, cholesterol, LDL, HDL, triglyceride, blood pressure, HbA1c, BMI, weight, waist circumference measurements will be evaluated. In this research, the exercise change stages dimension of the Transtheoretic Model will be discussed and the trainings will be planned according to these stages.

DETAILED DESCRIPTION:
11.1 Stages of Designing the Research

* The original English text of the Scale for Process of Exercise Engagement (SPEE), whose validity and reliability will be made, will be submitted for expert opinion and language translations will be made. In order to ensure language validity, reverse translation method will be used. For this, the scale will be translated from English to Turkish by three experts who know Turkish and English well and whose mother tongue is Turkish, and a joint Turkish translation will be created by the researchers. Later, the scale will be translated from Turkish to English by a different expert who does not know the original version of the scale.
* The Turkish form will be submitted to 10 faculty members for expert opinion in terms of content validity.
* The finalized scale will be applied to 20 patients who meet the criteria for inclusion in the sample group, and necessary arrangements will be made. The data of individuals with pre-application will not be used in the research.
* Validity and reliability studies of the finalized scale will be started.
* The study was planned to be carried out in family health centers located in the city center of Kilis. It was planned to include individuals diagnosed with prediabetes between the ages of 40 and 60 who volunteered to participate in the study, were able to perceive and answer questions, were literate, use mobile phones and read messages, have a smart phone, tablet or computer, have no problems with internet access, and were diagnosed with prediabetes.
* After the written consent form and informed consent form are obtained from the prediabetes patients who accepted to participate in the study, data will be collected for the validity-reliability of the scale.
* Prediabetes patients, who are invited to the family health center by phone by the researcher, will be taken to a suitable interview room where privacy will be ensured and a face-to-face form containing 40 questions in total, titled socio-demographic questions (10 questions), lifestyle behavior questions (15 questions), questions about co-morbid conditions (11 questions), questions about the use of health services (4 questions) will be filled by interview technique. The validity and reliability of the Scale for Process of Exercise Engagement (SPEE) (Turkish version) scale will be completed by the patients.
* After the determined number of data is collected, the steps necessary for the validity and reliability of the scale will be followed and the scale will be adapted to the Turkish society.
* For the second phase of the study, the Exercise Change Phase Short Questionnaire of the Transtheoretic Model and the Finnish Diabetes Risk Questionnaire (FINDRISK) will be applied to prediabetes patients who meet the research criteria. Individuals who get 14 points or more from the FINDRISK questionnaire and who are in the Not Thinking stage of the Exercise Change Phase Short Question Form will be determined and these individuals will be randomly assigned to the experimental and control groups. Pre-tests will be applied to the experimental and control groups. For the pre-test application, to the experimental and control groups; patient identification form (40 questions), Scale for Process of Exercise Engagement (SPEE) (Turkish version) will be applied as scale.
* At the beginning of the study, height measurements of the experimental and control groups will be made, body weights will be measured, and body mass indexes will be calculated and recorded. Their blood pressure will be measured and recorded.
* Blood samples will be taken to measure the fasting blood glucose, postprandial blood glucose, HgA1C, HDL, LDL, cholesterol and triglyceride values of the experimental and control groups and the results will be recorded in the metabolic values monitoring form.
* After the pre-tests, the exercise training and program, which was created as a result of the literature review, will be applied to the experimental group by videoconferencing method, taking into account the stages, processes and levels of the Transtheoretic Model. Training will be held via Zoom program. Each training will take approximately 40 minutes. The trainings will be once a week and a total of 5 weeks will be given and an exercise program will be applied. After each training, the 'Exercise Change Phase Short Question Form' of the Transtheoretic Model will be filled in again by the experimental group so that it will be checked at which stage of the change (not thinking, thinking, preparation, movement, maintaining) the patients are and the trainings will be arranged accordingly. Immediately after the training, the 'Exercise Change Phase of Transtheoretic Model' Short Question Form and Scale for Process of Exercise Engagement (SPEE) (Turkish version) will be applied to the experimental group, height and weight measurements will be made and recorded. Their blood pressure will be measured and recorded. Their blood tests will be taken and the results will be recorded in the metabolic values monitoring form.
* After the trainings are over, the experimental group will be followed up for 6 months in order to monitor the behavioral changes. During the follow-up phase, patients will be provided with the recommended exercise program. In the third month of the follow-up, the experimental and control groups will be asked to fill the Exercise Change Phase Short Question Form and Exercise Participation Process Scale, and their height, weight and blood pressure measurements will be made. Their HgA1C, HDL, LDL, triglyceride, cholesterol, fasting, postprandial blood sugars will be measured and recorded in the metabolic monitoring form. In addition, during this period, short messages created as a result of literature review will be sent to patients with prediabetes, taking into account the change stages, processes and levels of the Transtheoretic Model, 2 days a week, and the patients will be called once a week to answer their questions and motivate them to do the recommended exercises.
* After the preliminary test; The pedometer application will be downloaded to the smart mobile devices of the patients and the total number of daily steps of the patients will be calculated.
* The walking exercise follow-up book created by the researcher will be given to the patients after the pre-test. The purpose of the gait exercise follow-up book is to ensure the regular continuation of the patient's exercise program and to facilitate the follow-up of the patient. The patient will be asked to write the date, the time he/she started /finished walking, the number of steps and the complaints he/she encounters while walking, blood pressure, fasting and postprandial blood glucose values and weight measurements.
* No intervention or follow-up will be made to the control group in this process.
* In the posttest, the experimental and control groups will be provided to fill out the Exercise Change Phase Short Questionnaire of the Transtheoretic Model, the Finnish Diabetes Risk Questionnaire and the Exercise Participation Process Scale; their height and weight will be measured and their blood pressure will be checked and recorded. Their HgA1C, HDL, LDL, triglyceride, cholesterol, fasting, postprandial blood sugars will be measured and recorded in the metabolic monitoring form.
* After the posttest, an exercise training program based on the Transtheoretic Model will be given to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Individuals, diagnosed with prediabetes,
* 40-60 years old,
* A citizen of the Republic of Turkey,
* Not using drugs effective on blood glucose metabolism,
* No vision or hearing problems,
* No cognitive or psychiatric problems,
* Without diagnosis of malignancy,
* Not pregnant,
* Those who have a smartphone, tablet or computer, or a family member with devices with this feature, who have no problems with internet access,
* Able to use mobile phone and read messages,
* Residing in Kilis city center,
* Open to communication and cooperation,
* Literate,
* willing to participate in the study

Exclusion Criteria:

* Individuals who, don't have a smartphone, tablet, or computer, or don't have a family member with this feature,
* Having problems with internet access,
* are reluctant to participate in the study

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
The Effect of Health Education Given to Prediabetes Patients by Video Conferencing on Self-Management and Exercise Status | 6 months
  Among the metabolic control indicators of the traning group;
  * HbA1c value will be lower than the control group.
  * Cholesterol value will be lower than the control group.
  * LDL value will be lower than the control group
  * HDL value will be higher than the control group.
  * Triglyceride value will be lower than the control group.
The Effect of Health Education Given to Prediabetes Patients by Video Conferencing on Self-Management and Exercise Status | 6 months
  The blood pressure values (mmHg) of the group, who have been reminded by the health education given by video conferencing method and mobile communication tools, will be lower than the control group (manual sphygmomanometer).
The Effect of Health Education Given to Prediabetes Patients by Video Conferencing on Self-Management and Exercise Status | 6 months
  The weight (kg) of the group that has been reminded by the health education given by video conferencing method and mobile communication tools will be lower than the control group (Weighing instrument).
The Effect of Health Education Given to Prediabetes Patients by Video Conferencing on Self-Management and Exercise Status | 6 months
  BMI (kg/m2) of the group that has been reminded by the health education given by video conferencing method and mobile communication tools will be lower than the control group (Weighing instrument, height meter).
The Effect of Health Education Given to Prediabetes Patients by Video Conferencing on Self-Management and Exercise Status | 6 months
  Waist circumference (cm) of the group that has been reminded by the health education given by video conferencing method and mobile communication tools will be lower than the control group (tape measure).
The Effect of Health Education Given to Prediabetes Patients by Video Conferencing on Self-Management and Exercise Status | 6 months
  Compared to the control group, the mean score of participation developing awareness (min:4-max:20) will be higher for the group who have been reminded with health education given by video conferencing method and mobile communication tools Scale for Process of Exercise Engagement . Higher scores on the Developing Awareness (DA), represents higher levels for psychological and behavioral transitions, represents
The Effect of Health Education Given to Prediabetes Patients by Video Conferencing on Self-Management and Exercise Status | 6 months
  Compared to the control group, the mean score of participation creating the health blueprint (min:3-max:15) will be higher for the group who have been reminded with health education given by video conferencing method and mobile communication tools (Scale for Process of Exercise Engagement. Higher scores on the creating the health blueprint, represents higher levels for psychological and behavioral transitions, represents
The Effect of Health Education Given to Prediabetes Patients by Video Conferencing on Self-Management and Exercise Status | 6 months
  Compared to the control group, the mean score of participation driving force (min:6-max:30) will be higher for the group who have been reminded with health education given by video conferencing method and mobile communication tools Scale for Process of Exercise Engagement. Higher scores on the creating the driving force, represents higher levels for psychological and behavioral transitions, represents
The Effect of Health Education Given to Prediabetes Patients by Video Conferencing on Self-Management and Exercise Status | 6 months
  Compared to the control group, the mean score of participation spontaneous regular exercise (min:4-max20) will be higher for the group who have been reminded with health education given by video conferencing method and mobile communication tools (Scale for Process of Exercise Engagement. Higher scores on the creating the spontaneous regular exercise, represents higher levels for psychological and behavioral transitions, represents
The Effect of Health Education Given to Prediabetes Patients by Video Conferencing on Self-Management and Exercise Status | 6 months
  Compared to the control group, the mean score of participation resistive force (min: 4-max:20) will be lower for the group who have been reminded with health education given by video conferencing method and mobile communication tools (Scale for Process of Exercise Engagement. Higher scores on the creating the resistive force, represents lower levels for psychological and behavioral transitions, represents
The Effect of Health Education Given to Prediabetes Patients by Video Conferencing on Self-Management and Exercise Status | 6 months
  points (max:, min:) Developing awareness =4~20, Creating the health blueprint=3~15 Driving force= ,6~30 Resistive force= 4~20, Spontaneous regular exercise=4~20